CLINICAL TRIAL: NCT00775385
Title: Randomized Phase II/III Adjuvant Trial Evaluating Feasibility of Standard (A) vs. Customized Treatment (B) in Stage II or Stage IIIA Non-N2, Non-squamous Non Small Cell Lung Cancer (NSCLC).
Brief Title: TAilored Post-Surgical Therapy in Early Stage NSCLC
Acronym: TASTE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0801; Eudract : 2008-004939-38
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Chemotherapy, Adjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Standard chemotherapy
  Interventions: Drug: Standard Chemotherapy
- B (Experimental): Customized treatment
  Interventions: Drug: Customized Treatment

INTERVENTIONS:
Drug: Standard Chemotherapy — Pemetrexed Cisplatin Schedule : CDDP 75 mg/m² D1, pemetrexed 500 mg/m² D1 D1=D21, 4 cycles
  Arms: A
Drug: Customized Treatment — Mutated EGFR : Erlotinib 150mg/day (1 year)
  Wild-type EGFR or "undetermined" depends on ERCC1 status :
  * ERCC1 high : no treatment
  * ERCC1 low or undetermined : Pemetrexed Cisplatin, 4 cycles (63 days)
  Arms: B

SUMMARY:
Our hypothesis is that patients receiving therapy based on their baseline tumor ERCC1 levels and EGFR mutations would attain better disease free survival rates than patients in the control arm receiving noncustomized therapy. Using this selective approach, patients with stage II and IIIA non N2 NSCLC in the genotypic arm with low ERCC1 levels will receive cisplatin plus pemetrexed, and those with high ERCC1 levels will not receive cisplatin-based chemotherapy. If they harbor EGRF mutations they will be treated with erlotinib.

The study will be restricted to non-squamous NSCLC for two mains reasons. First, this will enrich the EGFR mutation rate that is awaited to be higher in these tumors than in squamous cell carcinoma. Second, permetrexed cisplatin combination has a promising efficacy and favorable toxicity profile and is of potential interest in the adjuvant setting of resected non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC that is defined as other than predominantly squamous cell histology (squamous cell and/or mixed small cell, non-small cell histology is not permitted)
* Surgically resected NSCLC with pathological stage II or stage IIIA non-N2 (TNM classification 2008)
* Performance status (PS) = 0 or 1
* 18 years <= age < 70 years
* Signed inform consent

Exclusion Criteria:

* Squamous cell carcinoma
* Previous cancer excepted those treated for more than 5 years and considered cured, basocellular skin carcinoma, carcinoma in situ of uterine cervix
* Inadequate renal or cardiac functions
* Pregnant women
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack, grade ≥ 2 peripheral neuropathy, peptic ulcer disease, erosive esophagitis or gastritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2016-01-21 (Actual)

PRIMARY OUTCOMES:
Feasibility (% of patients having started the treatment before 2 months after the surgery, with the biological results EGFR and ERCC1) | week

SECONDARY OUTCOMES:
Disease-free Survival | month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles SORIA, Pr, Principal Investigator — Institut Gustave Roussy (IGR); Marie Wislez, Pr, Principal Investigator — APHP - Hôpital Tenon (Paris)
Locations (42):
- France (42):
  - Centre Hospitalier, Aix-en-Provence
  - Clinique de L'Europe, Amiens
  - Angers - CHU, Angers
  - Centre Hospitalier, Béziers
  - Centre F. Baclesse, Caen
  - CHU - Pneumologie, Caen
  - Centre Hospitalier, Chauny
  - Chevilly Larue - CH, Chevilly-Larue
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - Clermont Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Dax - CH, Dax
  - Ermont - Clinique Claude Bernard, Ermont
  - CHU Grenoble - pneumologie, Grenoble
  - Le Mans - CHG, Le Mans
  - Centre Léon Bérard, Lyon
  - Lyon - Hôpital Louis Pradel (Pneumologie), Lyon
  - Mantes La Jolie - CH, Mantes-la-Jolie
  - APHM - Hôpital Sainte Marguerite, Marseille
  - Institut Paoli Calmette, Marseille
  - Metz - Belle Isle, Metz
  - Mont de Marsan - CH, Mont-de-Marsan
  - Montpellier - Clinique Clémentville, Montpellier
  - Mulhouse - CH, Mulhouse
  - Nancy - Polyclinique Gentilly, Nancy
  - Nevers - CH, Nevers
  - Paris - Saint Louis, Paris
  - APHP - Hopital Tenon - Pneumologie, Paris
  - Pau - CH, Pau
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Reims - CHU, Reims
  - Rennes - CHU, Rennes
  - Centre Hospitalier, Saint-Quentin
  - Nouvel Hopital Civil, Strasbourg
  - Hôpital Foch, Suresnes
  - Centre Hospitalier Intercommunal, Toulon
  - CHU Toulouse - Pneumologie, Toulouse
  - Clinique Pasteur, Toulouse
  - Tours - CHU, Tours
  - Nancy - CHU, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges

REFERENCES:
- [Result] Wislez M, Barlesi F, Besse B, Mazieres J, Merle P, Cadranel J, Audigier-Valette C, Moro-Sibilot D, Gautier-Felizot L, Goupil F, Renault A, Quoix E, Souquet PJ, Madroszyck A, Corre R, Perol D, Morin F, Zalcman G, Soria JC. Customized adjuvant phase II trial in patients with non-small-cell lung cancer: IFCT-0801 TASTE. J Clin Oncol. 2014 Apr 20;32(12):1256-61. doi: 10.1200/JCO.2013.53.1525. Epub 2014 Mar 17. PMID 24638013
- [Derived] Oudart JB, Garinet S, Leger C, Barlesi F, Mazieres J, Jeannin G, Audigier-Valette C, Morot-Sibilot D, Langlais A, Amour E, Mathiot N, Birsen G, Blons H, Wislez M. STK11/LKB1 alterations worsen the poor prognosis of KRAS mutated early-stage non-squamous non-small cell lung carcinoma, results based on the phase 2 IFCT TASTE trial. Lung Cancer. 2024 Apr;190:107508. doi: 10.1016/j.lungcan.2024.107508. Epub 2024 Feb 19. PMID 38428265
- See also: IFCT official website — http://www.ifct.fr